CLINICAL TRIAL: NCT06546449
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Escalating Doses of LH-001 in Healthy Participants
Brief Title: LH-001 vs Placebo in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chien-Liang Lin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Chien-Liang Lin, Professor of Neuroscience, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024W0061; 1U01AG068822-01 (NIH)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: LH-001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators and participants will remain blinded throughout the study. At the completion of each cohort, the statistician will be unblinded to analyze data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- SAD Cohort 1 (Experimental): Participants will be administered a single 12.5 mg dose of LH-001
  Interventions: Drug: LH-001
- SAD Cohort 2 (Experimental): Participants will be administered a single 25 mg dose of LH-001
  Interventions: Drug: LH-001
- SAD Cohort 3 (Experimental): Participants will be administered a single 50 mg dose of LH-001
  Interventions: Drug: LH-001
- SAD Cohort 4 (Experimental): Participants will be administered a single 100 mg dose of LH-001
  Interventions: Drug: LH-001
- MAD Cohort 1 (Experimental): Participants will be administered multiple 25 mg doses of LH-001
  Interventions: Drug: LH-001
- MAD Cohort 2 (Experimental): Participants will be administered multiple 50 mg doses of LH-001
  Interventions: Drug: LH-001
- MAD Cohort 3 (Experimental): Participants will be administered multiple 100 mg doses of LH-001
  Interventions: Drug: LH-001
- SAD Placebo cohorts 1, 2, 3 and 4 (Placebo Comparator): Participants will be administered a single dose of placebo
  Interventions: Drug: Placebo
- MAD Placebo cohorts 1, 2 and 3 (Placebo Comparator): Participants will be administered multiple doses of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LH-001 — LH-001 will be administered oral
  Arms: MAD Cohort 1; MAD Cohort 2; MAD Cohort 3; SAD Cohort 1; SAD Cohort 2; SAD Cohort 3; SAD Cohort 4
Drug: Placebo — Placebo will be administered oral
  Arms: MAD Placebo cohorts 1, 2 and 3; SAD Placebo cohorts 1, 2, 3 and 4

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of LH-001 when administered as an oral, single or multiple dose(s) at ascending dose levels in healthy participants.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, double-blinded, placebo-controlled study. This study consists of two parts: (1) single ascending doses in 4 cohorts (SAD) and (2) 14-day multiple ascending doses in 3 cohorts (MAD). Cohorts may be added or removed if needed due to safety considerations or deviations of actual PK parameters from predicted values.

The SAD study consists of a screening visit, a 2-day inpatient stay (Day 1-2), a return visit for safety assessments on Day 3, Day 4, and Day 8.

The MAD study consists of a screening visit, a 2-day inpatient stay (Day 1-2), daily return for dosing and safety assessments (Day 3-13), a 2-day inpatient stay (Day 14-15), and a follow-up by phone (Day 21).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-60 years at the time of consent
* Must provide written informed consent
* Physically and mentally able and willing to participate in the safety and other assessments including staying overnight
* BMI 18-29.9 kg/m2
* Sexually active male participants, sexually active female participants of childbearing potential, and their sexual partners are to adhere to the contraception requirements. These requirements include utilizing highly effective birth control (including hormonal methods, intrauterine devices, and/or barrier methods) from the screening phase through the completion of the last study follow-up. Note, the barrier method may not be used as a standalone method and must be combined with an additional approved method.
* Participants taking non-prescribed medication must cease taking the medication for at least 48 hours prior to dosing of LH-001.

Exclusion Criteria:

* Taking any prescription medications outlined in the prohibited/conditional drug list (see Section 6.8.1)
* History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History or presence of major disorder of any other major organ system (cardiovascular, respiratory, central nervous system, or endocrine system)
* History of cancer within 5 years of consent (exceptions are squamous and basal cell carcinomas of the skin)
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dosing.
* History or presence of alcohol or substance abuse
* History of chronic or current use of recreational or illicit drugs
* History of, or treatment for, major psychiatric illness
* History of, or treatment for, seizures or epilepsy
* Pregnant or breast-feeding females
* History of, or treatment for, an autoimmune disease (e.g., Rheumatoid Arthritis, Multiple Sclerosis, Myasthenia Gravis, etc.)
* History of asplenia, hyposplenia, or splenectomy
* History or presence of drug hypersensitivity
* Poor venous access
* Receipt of investigational therapy within 4 months prior to screening
* Current or previous use of systemic corticosteroids or other systemic immunosuppressive agents 4 weeks prior to dosing
* Current or previous use of NMDA antagonists 4 weeks prior to dosing
* Clinically significant findings in the opinion of the investigator in the laboratory, physical examination, or vital sign assessments
* Evidence of active Hepatitis B, Hepatitis C, or HIV on laboratory testing
* Any clinically significant ECG abnormality in the opinion of the investigator
* Plasma or blood donation within the last 4 weeks
* Positive drug or alcohol screen
* Any contraindication to or unable to tolerate a LP, for those who consented to the procedure, including the use of anti-coagulant medications. Daily administration of 81 mg aspirin will be allowed
* Any concurrent condition that, in the opinion of the investigator, would interfere with the evaluation of LH-001
* Participants who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this CSSRS Item 5 occurred within the last 6 months OR Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred in the last 2 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who experience at least one treatment-emergent AE | 8 days for SAD and 21 days for MAD
Percentage of participants who discontinue due to an AE | 8 days for SAD and 21 days for MAD
Percentage of participants who meet the markedly abnormal criteria for vital sign measurements at least once post-dose | 8 days for SAD and 21 days for MAD
Percentage of participants who meet the markedly abnormal criteria for safety ECG parameters at least once post-dose | 8 days for SAD and 21 days for MAD
Percentage of participants who meet the markedly abnormal criteria for safety laboratory tests at least once post-dose | 8 days for SAD and 21 days for MAD

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Day 1 for all cohorts and Day 14 for MAD cohorts
Time to reach maximum concentration (Tmax) | Day 1 for all cohorts and Day 14 for MAD cohorts
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration (AUC0-last) | Day 1 for all cohorts and Day 14 for MAD cohorts
Time for LH-001 concentration to fall to half of its original value (T½) | Day 1 for all cohorts and Day 14 for MAD cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Liang Glenn Lin, PhD, Study Director — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No